CLINICAL TRIAL: NCT00876421
Title: A Randomised, Multi-Centre, Double-Blind, Placebo and Active-Controlled, 5-Way Parallel Group Study to Investigate the Efficacy, Safety and Tolerability of ONO-8539 in Patients With Overactive Bladder
Brief Title: Study of ONO-8539 in Patients With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-8539POE004
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Overactive Bladder
Keywords: ONO-8539; Overactive bladder; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; ONO-8539

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- P (Placebo Comparator)
  Interventions: Drug: Placebo
- A (Active Comparator)
  Interventions: Drug: Tolterodine
- E1 (Experimental)
  Interventions: Drug: ONO-8539
- E2 (Experimental)
  Interventions: Drug: ONO-8539
- E3 (Experimental)
  Interventions: Drug: ONO-8539

INTERVENTIONS:
Drug: Placebo — Placebo / 12 weeks
  Arms: P
Drug: Tolterodine — 4mg / 12 weeks
  Arms: A
Drug: ONO-8539 — low dose / 12 weeks
  Arms: E1
Drug: ONO-8539 — medium dose / 12 weeks
  Arms: E2
Drug: ONO-8539 — higher dose / 12 weeks
  Arms: E3

SUMMARY:
The objective of this study is to investigate efficacy, safety and tolerability of ONO-8539 in patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical history of Overactive Bladder symptoms for > 6 months

Exclusion Criteria:

* Patients who have a history or presence of other significant diseases, which in the opinion of the investigator, might compromise the patient's safety or the evaluation of the study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Overactive bladder symptoms | 12 weeks

SECONDARY OUTCOMES:
Overactive bladder symptoms (QOL) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Kuwayama, Study Director — Clinical Development, ONO Pharma UK, Ltd
Locations (50):
- Czechia (8):
  - Brno
  - Jindřichův Hradec
  - Olomouc
  - Opava
  - Pilsen
  - Prague
  - Štětí
  - Ústí nad Labem
- Germany (6):
  - Duisburg
  - Hagenow
  - Krumbach
  - Magdeburg
  - Mülheim
  - Weiden
- Hungary (5):
  - Budapest
  - Dombóvár
  - Nyíregyháza
  - Szeged
  - Szekszárd
- Netherlands (5):
  - Heerlen
  - Maastricht
  - The Hague
  - Tilburg
  - Winterswijk
- Poland (9):
  - Bialystok
  - Bielsko-Biala
  - Gdansk
  - Gdynia
  - Katowice
  - Lodz
  - Lublin
  - Mysłowice
  - Warsaw
- Romania (4):
  - Arad
  - Bihor
  - Bucharest
  - Timuș
- Russia (3):
  - Moscow
  - Rostov-on-Don
  - Saint Petersburg
- Sweden (5):
  - Gothenburg
  - Kungälv
  - Stockholm
  - Umeå
  - Uppsala
- Ukraine (5):
  - Chernivtsi
  - Donetsk
  - Kharkiv
  - Kyiv
  - Zaporizhzhya